CLINICAL TRIAL: NCT06167096
Title: Effects of Lavender Aromatherapy on Patient Anxiety During Mohs Micrographic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE8Z23
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Skin Cancer; Skin Carcinoma
Keywords: Skin Cancer; Lavender Aromatherapy
MeSH Terms: conditions — Skin Neoplasms | interventions — lavender oil; Water

STUDY DESIGN:
Intervention Model Description: This study is a single-blinded randomized control study. Days before surgery, participants meeting inclusion criteria will be contacted and an electronic consent will be completed. The intervention shall not be disclosed to participants. Days in which lavender is used in clinic will alternate; participants will be scheduled as normal. participants will therefore be randomly assigned to one of two groups, lavender or control, depending on their surgery date. On the day of surgery, participants who previously completed the electronic consent will be brought to a room with a diffuser. The diffusers will be turned on 15 minutes before scheduled time of surgery with lavender for the intervention group (4 drops per 100ml water) or just water for the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender (Experimental): 4 drops of lavender essential oil will be added to an electronic diffusion device with 100ml of water. The device will be turned on 15 minutes before surgery for participants who previously agreed to the study. The device will be turned off after completion of the post- layer questionnaires assessing anxiety and participant experience.
  Interventions: Other: Lavender essential oil
- Water (Placebo Comparator): On the day of surgery, participants who previously completed the electronic consent will be brought to a room with a diffuser. The diffusers will be turned on 15 minutes before scheduled time of surgery with just water for the control group
  Interventions: Other: Water

INTERVENTIONS:
Other: Lavender essential oil — Lavender Oil; blend of two (2) pure lavender oil - Lavandula angustifolia from Bulgaria and Lavandula hybrida from France
  Arms: Lavender
Other: Water — Water
  Arms: Water

SUMMARY:
This study aims to improve patient comfort by exploring the potential of lavender aromatherapy in reducing anxiety and unpleasant odor perception during Mohs Micrographic Surgery (MMS).

Lavender has been widely studied for its sedative-like properties and calming effects, both in medical and dental settings. By investigating the impact of lavender aromatherapy on patient anxiety levels during MMS, we seek to provide evidence-based insights into non- pharmacological interventions that can enhance the overall comfort and experience of participants.

DETAILED DESCRIPTION:
Mohs Micrographic Surgery (MMS) is a precise and highly effective technique used to treat skin cancers, particularly those with complex or recurrent features. Despite its proven clinical benefits, MMS can be an anxiety-inducing experience for some participants, attributed to the anticipation of the procedure, potential postoperative pain, and the perception of unpleasant odors during the surgical stages; nearly 66% of participants undergoing MMS report unpleasant smells. Anxiety has been shown to adversely affect participants' postoperative recovery and may heighten the perception of pain.

Traditional interventions to manage anxiety in medical settings often involve medication, which may not align with patient preferences. Therefore, there is a need to explore alternative non-pharmacological approaches to create a calming environment during MMS. One such promising intervention is the use of lavender aromatherapy, known for its sedative-like properties and calming effects in various settings. A growing body of research supports the potential benefits of lavender in promoting relaxation and reducing anxiety. Studies conducted on animal models have demonstrated lavender's sedative-like properties, and its active component, linalool, has been shown to inhibit limbic system activity and decrease sympathetic nerve activity.

The inhalation of lavender aroma has been found to influence brain activity, resulting in increased carbohydrates and decreased neurotransmitter activity. Moreover, lavender oil has also been widely studied in dental literature, where it has demonstrated remarkable potential in reducing patient anxiety during various dental procedures.

Another non-pharmacological intervention commonly used to alleviate patient anxiety is music. Music during MMS leads to significant decreases in patient reported anxiety levels, as well as physiological indicators of anxiety. Patient selected music leads to an even greater reduction in anxiety. Despite the positive findings in various medical settings, there is a notable gap in research regarding the application of lavender aromatherapy during MMS and its impact on anxiety levels and unpleasant odor perception. This research aims to investigate the potential of lavender aromatherapy in promoting a calming environment during MMS and its effects on reducing anxiety levels and the perception of unpleasant smells. The study will explore how lavender diffuser use in operating rooms influences patient anxiety levels during the surgical process. By examining the experiences of participants undergoing MMS, this study seeks to provide valuable insights into the efficacy of non-pharmacological interventions, particularly aromatherapy, in reducing anxiety levels and enhancing the overall patient experience during MMS. The findings could contribute to the development of evidence-based interventions to alleviate patient anxiety and improve the overall surgical process for those undergoing MMS

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* No previous Mohs surgeries
* Currently seen in UH(University Hospitals)Westlake Dermatology Clinic for Mohs surgery
* Mohs surgery of the head and neck

Exclusion Criteria:

* Participants with lavender allergies
* Participants with aroma sensitivities
* Participants with anosmia
* Participants with cold or flu symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in participant anxiety levels as measured by STAI assessment scale | Before MMS procedure
  Anxiety levels will be measured using the 6-question Spielberg State Trait Anxiety Inventory (STAI) with scale from 1-4, 1 being low and 4 being high
Change in participant anxiety levels as measured by STAI assessment scale | After MMS procedure post 1 layer
  Anxiety levels will be measured using the 6-question Spielberg State Trait Anxiety Inventory (STAI) with scale from 1-4, 1 being low and 4 being high
Change in participant anxiety levels as measured by VAS assessment scale | Before MMS procedure
  Anxiety levels will be measured using Visual Analog Scale (VAS) of 0 to 100 where 0 being calm and 100 being anxious
Change in participant anxiety levels as measured by VAS assessment scale | After MMS procedure post 1 layer
  Anxiety levels will be measured using Visual Analog Scale (VAS) of 0 to 100 where 0 being calm and 100 being anxious

SECONDARY OUTCOMES:
Perception of unpleasant smells | After MMS procedure post 1 layer
  Perception of unpleasant smells will be assessed using a participant satisfaction survey administered post-1 layer with a scale from 0 to 10, 0 being rated as poor/week and 10 being rated as excellent/strong

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Carroll, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No